CLINICAL TRIAL: NCT00604396
Title: Safety and Efficacy of Insulin Detemir Combined With OAD Versus Insulin NPH Combined With OAD in Type 2 Mellitus
Brief Title: Safety and Efficacy of Insulin Detemir in Combination With OAD in Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN304-1530
Record Dates: First submitted 2008-01-17; First posted 2008-01-30 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Insulin Detemir; Insulin, Isophane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: insulin detemir
Drug: insulin NPH

SUMMARY:
This trial is conducted in Europe.

The aim of this trial is to investigate the safety and efficacy of insulin detemir combined with oral anti-diabetic drugs (OADs) versus insulin NPH combined with oral anti-diabetic drugs (OADs) in Type 2 mellitus not well controlled on current therapy on blood glucose control.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes for at least 12 months since diagnosis
* Insulin naive subjects
* OAD treatment for at least 4 months alone or combined with no more than two OADs
* Body mass index (BMI) below 35.0 kg/m2
* HbA1c between 7.5-10.0%
* Able and willing to use twice a day injections for the entire trial period

Exclusion Criteria:

* Current or previous treatment with thiazolidiones within the last 6 months
* OAD treatment with three or more OADs within the last 6 months
* Acute insulin treatment for longer than 7 days in a row within the last 6 months
* Secondary diabetes
* Known maturity onset of diabetes of young (MODY)
* Known or suspected allergy to trial product or related products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 477 (Actual)
Dates: Start 2003-03; Primary Completion 2004-01 (Actual); Study Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
HbA1c | after 26 weeks of treatment

SECONDARY OUTCOMES:
Fasting plasma glucose
Within-subject variation
Incidence of total hypoglycaemic episodes
Body weight
Incidence of adverse events
Insulin antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (55):
- Belgium (4):
  - Novo Nordisk Investigational Site, Arlon
  - Novo Nordisk Investigational Site, Gilly
  - Novo Nordisk Investigational Site, Huy
  - Novo Nordisk Investigational Site, Jumet
- Croatia (2):
  - Novo Nordisk Investigational Site, Rijeka
  - Novo Nordisk Investigational Site, Zagreb
- Denmark (8):
  - Novo Nordisk Investigational Site, Århus C
  - Novo Nordisk Investigational Site, Copenhagen
  - Novo Nordisk Investigational Site, Hjørring
  - Novo Nordisk Investigational Site, Hvidovre
  - Novo Nordisk Investigational Site, Kalundborg
  - Novo Nordisk Investigational Site, København S
  - Novo Nordisk Investigational Site, Køge
  - Novo Nordisk Investigational Site, Slagelse
- France (11):
  - Novo Nordisk Investigational Site, Amiens
  - Novo Nordisk Investigational Site, Auxerre
  - Novo Nordisk Investigational Site, Avignon
  - Novo Nordisk Investigational Site, Dax
  - Novo Nordisk Investigational Site, Évry
  - Novo Nordisk Investigational Site, Mougins
  - Novo Nordisk Investigational Site, Nanterre
  - Novo Nordisk Investigational Site, Nevers
  - Novo Nordisk Investigational Site, Rueil-Malmaison
  - Novo Nordisk Investigational Site, Valenciennes
  - Novo Nordisk Investigational Site, Vénissieux
- Novo Nordisk Investigational Site, Skopje, North Macedonia
- Norway (9):
  - Novo Nordisk Investigational Site, Bekkestua
  - Novo Nordisk Investigational Site, Bergen
  - Novo Nordisk Investigational Site, Elverum
  - Novo Nordisk Investigational Site, Gjettum
  - Novo Nordisk Investigational Site, Gjøvik
  - Novo Nordisk Investigational Site, Jessheim
  - Novo Nordisk Investigational Site, Oslo
  - Novo Nordisk Investigational Site, Rådal
  - Novo Nordisk Investigational Site, Stavanger
- Poland (10):
  - Novo Nordisk Investigational Site, Gniewkowo
  - Novo Nordisk Investigational Site, Krakow
  - Novo Nordisk Investigational Site, Lodz
  - Novo Nordisk Investigational Site, Lublin
  - Novo Nordisk Investigational Site, Rawa Mazowiecka
  - Novo Nordisk Investigational Site, Szczecin
  - Novo Nordisk Investigational Site, Tychy
  - Novo Nordisk Investigational Site, Warsaw
  - Novo Nordisk Investigational Site, Wołomin
  - Novo Nordisk Investigational Site, Zabrze
- Russia (2):
  - Novo Nordisk Investigational Site, Moscow
  - Novo Nordisk Investigational Site, Saint Petersburg
- Novo Nordisk Investigational Site, Trenčín, Slovakia
- Sweden (7):
  - Novo Nordisk Investigational Site, Falun
  - Novo Nordisk Investigational Site, Grästorp
  - Novo Nordisk Investigational Site, Kristianstad
  - Novo Nordisk Investigational Site, Linköping
  - Novo Nordisk Investigational Site, Lund
  - Novo Nordisk Investigational Site, Trelleborg
  - Novo Nordisk Investigational Site, Umeå

REFERENCES:
- [Result] Hermansen K, Davies M, Derezinski T, Martinez Ravn G, Clauson P, Home P. A 26-week, randomized, parallel, treat-to-target trial comparing insulin detemir with NPH insulin as add-on therapy to oral glucose-lowering drugs in insulin-naive people with type 2 diabetes. Diabetes Care. 2006 Jun;29(6):1269-74. doi: 10.2337/dc05-1365. PMID 16732007
- [Result] Davies MJ, Derezinski T, Pedersen CB, Clauson P. Reduced weight gain with insulin detemir compared to NPH insulin is not explained by a reduction in hypoglycemia. Diabetes Technol Ther. 2008 Aug;10(4):273-7. doi: 10.1089/dia.2008.0282. PMID 18715200
- [Derived] Semlitsch T, Engler J, Siebenhofer A, Jeitler K, Berghold A, Horvath K. (Ultra-)long-acting insulin analogues versus NPH insulin (human isophane insulin) for adults with type 2 diabetes mellitus. Cochrane Database Syst Rev. 2020 Nov 9;11(11):CD005613. doi: 10.1002/14651858.CD005613.pub4. PMID 33166419
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com